CLINICAL TRIAL: NCT05487417
Title: Effects of Minocycline on Patients With Acute Anterior Circulation Ischemic Stroke Undergoing Intravenous Thrombectomy
Brief Title: Effects of Minocycline on Patients With Ischemic Stroke Undergoing Intravenous Thrombectomy
Acronym: MIST-A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Xi'an No.3 Hospital (Other Government); Xi'an Gaoxin Hospital (Other); First People's Hospital of Xianyang (Other); Xi'an XD Group Hospital (Unknown); Baoji High-tech Hospital (Unknown); Weinan Central Hospital (Other); Xi'An Daxing Hospital (Unknown); Yan'an University Xianyang Hospital (Unknown); The First Hospital of Yulin (Unknown); Northwest University First Hospital (Unknown); Jingyang County Hospital (Unknown); Yulin No.2 Hospital (Other); Yan'an people's Hospital (Unknown); Yuncheng Central Hospital (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Xi'an No.9 Hospital (Unknown); First Affiliated Hospital Xi'an Jiaotong University (Other); Pucheng County Hospital (Unknown)
Responsible Party: Principal Investigator, Wen Jiang-3, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJLL-KY20222186
Record Dates: First submitted 2022-07-30; First posted 2022-08-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Minocycline; Mechanical thrombectomy; Anterior circulation; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the outcome of minocycline group and routine treatment group was compared. Placebo control was not used, so outcomes assessor blind was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline treatment group (Experimental): Patients were given minocycline 200mg/d orally from the day of admission for 5 days. At the same time, the patient received mechanical thrombectomy and other standard treatments for acute ischemic stroke.
  Interventions: Drug: Minocycline
- Routine treatment group (No Intervention): Patients were given mechanical thrombectomy and other standard treatment for acute ischemic stroke, without minocycline treatment.

INTERVENTIONS:
Drug: Minocycline — Minocycline is a tetracycline antibiotic. Previous studies have confirmed that its application in stroke patients has good efficacy and safety, suggesting that it could become a synergistic treatment of mechanical thrombectomy.
  Arms: Minocycline treatment group

SUMMARY:
Minocycline is the second generation of tetracycline. Because of its lipophilicity, it has high penetrance of blood-brain barrier. Animal model studies have shown that minocycline can reduce cerebral damage after ischemic stroke, and its mechanism involves multiple molecular pathways, such as antioxidant, anti-inflammatory, anti apoptotic pathways, and protection of blood-brain barrier. Clinical studies have also shown that minocycline can significantly improve 3-month National Institute of Health Stroke Scale (NIHSS) and modified Rankin Scale (mRS) of patients with ischemic stroke, indicating that minocycline is a potential neuroprotective drug. Minocycline is believed to protect the blood-brain barrier, thereby reducing the ischemia-reperfusion injury caused by mechanical thrombectomy. However, whether minocycline can become a synergistic treatment method of mechanical thrombectomy, there is no clinical research in this area at present. Therefore, investigators carry out the study on the effect of minocycline in patients with acute anterior circulation ischemic stroke after mechanical thrombectomy, and plan to enroll 180 patients. To explore the safety and effectiveness of minocycline in patients with acute ischemic stroke after thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute cerebral infarction of anterior circulation accompanied by large vessel occlusion;
2. Age 18-85 years old;
3. The time of onset ≤ 6 hours or ≤ 24 hours suitable for mechanical thrombectomy determined by multimodal imaging;
4. The time of onset 6-24 hours, DWI shows an infarct volume less than 1/3 of the MCA blood supply area; the time of onset ≤ 6 hours, the ASPECTS(Alberta Stroke Program Early CT Score) is ≥6;
5. Preoperative NIHSS score ranges from 6 to 30 points;
6. Sign the informed consent form;

Exclusion Criteria:

1. There are contraindications for mechanical thrombectomy;
2. No revascularization therapy was performed during the operation or the TICI score after revascularization therapy was less than 2b;
3. There are other major central nervous system diseases, such as brain injury, brain tumor, multiple sclerosis, etc;
4. There is evidence that the patient has bacterial endocarditis, aortic dissection, arteritis or venous cerebral infarction;
5. Renal insufficiency or hepatic insufficiency (serum creatinine >2.0 mg/dL or 180 µmol/L; liver function greater than 3 times the normal value);
6. Known history of congestive heart failure (requiring dietary or medication changes or hospitalization) within 6 months, or myocardial infarction within 6 months;
7. There is evidence of any other life-threatening or severe diseases that may hinder the completion of the 3-month follow-up and affect the evaluation of the results;
8. Pre-existing neurological deficits or history of dementia;
9. There are infectious diseases that require antibiotic treatment before the disease;
10. Allergic to tetracyclines or unable to take minocycline for other reasons;
11. Minocycline could not be given within 1 hour after recanalization;
12. Pregnant patients;
13. Participated in another clinical trial within 30 days before inclusion in the study.
14. Refuse to sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in infarct volume from baseline to day 5 | Day 5 after onset
  Baseline infarct volume is measured by diffusion-weighted imaging (DWI), day 5 infarct volume is measured by fluid attenuated inversion recovery (FLAIR), Images are processed by imSTROKE software.

SECONDARY OUTCOMES:
Functional outcome at 3 months after onset | 3 months after onset
  Defined by the modified Rankin Scale (mRS), which ranges from 0 (no symptoms) to 6 (death), analyzed for superiority and then for noninferiority.
Favourable outcome at 3 months after onset | 3 months after onset
  Defined as proportion of patients with modified Rankin Scale (mRS) 0-2, which ranges from 0 (no symptoms) to 6 (death), An mRS score of <3 indicated a favourable outcome, whereas a score of ≥3 indicated a poor outcome.
Excellent outcome at 3 months after onset | 3 months after onset
  Defined as proportion of patients with modified Rankin Scale (mRS) 0-1, which ranges from 0 (no symptoms) to 6 (death), An mRS score of <2 indicated a excellent outcome, whereas a score of ≥2 indicated a poor outcome.
Improvement of neurological function compared with baseline | day 1, day 3, day 5, day 7, and 3 months after onset
  Defined by the National Institute of Health Stroke Scale (NIHSS), which ranges from 0 (no neurological injury) to 42 (severe neurological injury). The assessment time points were baseline, day 1, day 3, day 5, day 7, and 3 months after onset.
Improvement of activity of daily living at 3 months after onset | 3 months after onset
  Defined by Barthel index (BI), which ranges from 0 (completely lose the ability to live independently) to 100 (complete ability to live independently). The assessment time points were 3 months after onset
Incidence of intracranial hemorrhage at day 1 after onset | Day 1 after onset
  Intracranial hemorrhage is measured by CT scan. Images are processed by RAPID ICH software.
Mortality at 3 months after onset | 3 months after onset
  The investigators record all-cause mortality
Infarct volume at day 5 after onset | Day 5 after onset
  Day 5 infarct volume is measured by fluid attenuated inversion recovery (FLAIR). Images are processed by imSTROKE software.
Length of hospital stay and length of Intensive Care Unit (ICU) stay | 3 months after onset
  How long the patients stay in hospital, and how long the patients stay in ICU

OTHER OUTCOMES:
Safety outcomes: adverse events and serious adverse events | 3 months after onset
  Safety outcomes were incidences of adverse events and serious adverse events that were related or not related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Background] Yenari MA, Xu L, Tang XN, Qiao Y, Giffard RG. Microglia potentiate damage to blood-brain barrier constituents: improvement by minocycline in vivo and in vitro. Stroke. 2006 Apr;37(4):1087-93. doi: 10.1161/01.STR.0000206281.77178.ac. Epub 2006 Feb 23. PMID 16497985
- [Background] Matsukawa N, Yasuhara T, Hara K, Xu L, Maki M, Yu G, Kaneko Y, Ojika K, Hess DC, Borlongan CV. Therapeutic targets and limits of minocycline neuroprotection in experimental ischemic stroke. BMC Neurosci. 2009 Oct 6;10:126. doi: 10.1186/1471-2202-10-126. PMID 19807907
- [Background] Liao TV, Forehand CC, Hess DC, Fagan SC. Minocycline repurposing in critical illness: focus on stroke. Curr Top Med Chem. 2013;13(18):2283-90. doi: 10.2174/15680266113136660160. PMID 24059465
- [Background] Yang Y, Salayandia VM, Thompson JF, Yang LY, Estrada EY, Yang Y. Attenuation of acute stroke injury in rat brain by minocycline promotes blood-brain barrier remodeling and alternative microglia/macrophage activation during recovery. J Neuroinflammation. 2015 Feb 10;12:26. doi: 10.1186/s12974-015-0245-4. PMID 25889169
- [Background] Muhammad S, Planz O, Schwaninger M. Increased Plasma Matrix Metalloproteinase-9 Levels Contribute to Intracerebral Hemorrhage during Thrombolysis after Concomitant Stroke and Influenza Infection. Cerebrovasc Dis Extra. 2016;6(2):50-9. doi: 10.1159/000447750. Epub 2016 Aug 25. PMID 27560521
- [Background] Fagan SC, Waller JL, Nichols FT, Edwards DJ, Pettigrew LC, Clark WM, Hall CE, Switzer JA, Ergul A, Hess DC. Minocycline to improve neurologic outcome in stroke (MINOS): a dose-finding study. Stroke. 2010 Oct;41(10):2283-7. doi: 10.1161/STROKEAHA.110.582601. Epub 2010 Aug 12. PMID 20705929
- [Background] Lampl Y, Boaz M, Gilad R, Lorberboym M, Dabby R, Rapoport A, Anca-Hershkowitz M, Sadeh M. Minocycline treatment in acute stroke: an open-label, evaluator-blinded study. Neurology. 2007 Oct 2;69(14):1404-10. doi: 10.1212/01.wnl.0000277487.04281.db. PMID 17909152
- [Background] Elkins J, Veltkamp R, Montaner J, Johnston SC, Singhal AB, Becker K, Lansberg MG, Tang W, Chang I, Muralidharan K, Gheuens S, Mehta L, Elkind MSV. Safety and efficacy of natalizumab in patients with acute ischaemic stroke (ACTION): a randomised, placebo-controlled, double-blind phase 2 trial. Lancet Neurol. 2017 Mar;16(3):217-226. doi: 10.1016/S1474-4422(16)30357-X. Epub 2017 Feb 15. PMID 28229893
- [Background] Nogueira RG, Jadhav AP, Haussen DC, Bonafe A, Budzik RF, Bhuva P, Yavagal DR, Ribo M, Cognard C, Hanel RA, Sila CA, Hassan AE, Millan M, Levy EI, Mitchell P, Chen M, English JD, Shah QA, Silver FL, Pereira VM, Mehta BP, Baxter BW, Abraham MG, Cardona P, Veznedaroglu E, Hellinger FR, Feng L, Kirmani JF, Lopes DK, Jankowitz BT, Frankel MR, Costalat V, Vora NA, Yoo AJ, Malik AM, Furlan AJ, Rubiera M, Aghaebrahim A, Olivot JM, Tekle WG, Shields R, Graves T, Lewis RJ, Smith WS, Liebeskind DS, Saver JL, Jovin TG; DAWN Trial Investigators. Thrombectomy 6 to 24 Hours after Stroke with a Mismatch between Deficit and Infarct. N Engl J Med. 2018 Jan 4;378(1):11-21. doi: 10.1056/NEJMoa1706442. Epub 2017 Nov 11. PMID 29129157
- [Derived] Zhang X, Zhao J, Sun Z, Wei D, Yao L, Li W, Zhu H, Liu W, Zhang H, Yuan X, Ma X, Meng J, Wang B, Jia Y, Qin N, Jiang W; MIST-A Study Group. Effects of minocycline on patients with acute anterior circulation ischaemic stroke undergoing intravenous thrombectomy (MIST-A): the study protocol for a multicentre, prospective, randomised, open-label, blinded-endpoint trial. BMJ Open. 2024 Dec 20;14(12):e093443. doi: 10.1136/bmjopen-2024-093443. PMID 39806586